CLINICAL TRIAL: NCT04306003
Title: Enhanced Recovery After Surgery in Autologous Breast Reconstruction: A Pilot Randomized Controlled Trial
Brief Title: ERAS in Autologous Breast Reconstruction: A Pilot RCT
Acronym: ERAS-ABR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Brian Hyosuk Chin, Principal Investigator, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERAS-ABR
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Reconstruction; Perioperative Care; Enhanced Recovery After Surgery; ERAS
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: ERAS is a complex intervention in which care providers cannot be blinded. Patients were provided a brief overview of ERAS without specific details of its interventions but were not informed of the group allocation. Patients were unaware of group allocation as they were unaware of the specific differences in the perioperative care between ERAS and standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Recovery After Surgery (ERAS) pathway (Experimental): Preop
  1. Diet: Solids until midnight before surgery with a carbohydrate rich drink before midnight and 3-hours prior to surgery.
  2. Analgesia: Acetaminophen 975mg & Celecoxib 400mg administered PO 1-hour before surgery.
  Intraop
  1. Hypothermia prevention: Forced-air warming units and core temperature monitoring.
  2. Fluid management: Euvolemic fluid management with balanced crystalloid solution.
  3. Analgesia: 0.25% bupivacaine block of intercostal nerves and rectus sheath by the surgical team. Additional IV analgesia by anesthesiologist with the goal to minimize opioids.
  4. PONV prophylaxis: Ondansetron 4-8mg IV during emergence.
  Postop
  1. Diet: Clear fluids immediately post-op. Saline lock and advance to DAT on POD#1.
  2. Analgesia: Routine administration of Acetaminophen 975mg PO q6h & Celecoxib 200mg PO q12h. Opioids used as breakthrough analgesia only. No PCA.
  3. Early mobilization: Mobilization within the first 24 hours after surgery with assistance.
  Interventions: Other: ERAS pathway
- Standard Perioperative Care (Active Comparator): Patients in the control arm received routine perioperative care as determined by respective surgeons participating in the study.
  Interventions: Other: Standard Perioperative Care

INTERVENTIONS:
Other: ERAS pathway — See ERAS pathway arm description.
  Arms: Enhanced Recovery After Surgery (ERAS) pathway
Other: Standard Perioperative Care — See control arm description.
  Arms: Standard Perioperative Care

SUMMARY:
Over 26,000 Canadian women are diagnosed with breast cancer each year and 1 in 3 patients undergo mastectomy. With an upward of 40% of breast cancer patients seeking post-mastectomy breast reconstruction (PMBR), there is a significant opportunity to improve the quality of perioperative care for breast reconstruction patients. Enhanced Recovery After Surgery (ERAS) is a multidisciplinary, multimodal, and evidence-based approach to perioperative care that safely reduces hospital length of stay and opioid use following colorectal surgery. ERAS recommendations have been proposed for women undergoing autologous PMBR who typically stay in hospital 4 to 5 days after surgery. However, the evidence to support ERAS in breast reconstruction is limited to observational studies compared to the numerous clinical trials in colorectal surgery. The goal of this study is to address this knowledge gap by evaluating the feasibility of conducting a RCT comparing ERAS to standard perioperative care.

DETAILED DESCRIPTION:
1.1 Primary research question To determine the feasibility of a randomized controlled trial comparing an Enhanced Recovery After Surgery (ERAS) protocol to conventional perioperative care for adult women with breast cancer undergoing post-mastectomy autologous breast reconstruction.

1.2 Background and rationale Over 26,000 Canadian women are diagnosed with breast cancer every year. While the 5-year survival of breast cancer has improved to 87% in Canada, 1 in 3 breast cancer patients that receive mastectomy experience a negative impact in quality of life. Breast reconstruction can improve the physical, psychosocial and sexual well-being of patients after mastectomy. With an upward of 40% of breast cancer patients who undergo post-mastectomy breast reconstruction, there is a significant opportunity to improve the quality of surgical care for breast reconstruction patients.

Breast reconstruction can be classified into alloplastic (implant-based) and autologous (tissue-based) reconstruction. While alloplastic reconstruction is the most common form of breast reconstruction in North America, autologous reconstruction using the patient's own tissue confers superior long-term satisfaction and quality of life. The gold standard of autologous reconstruction is the deep inferior epigastric perforator (DIEP) flap which uses the patients' abdominal tissue to reconstruct the breast using microvascular techniques, while preserving the abdominal musculature. The DIEP reconstruction is surgically more complex than the alloplastic approach, involving surgery at the breasts, abdominal donor site, and reattachment of the abdominal tissue to blood vessels in the chest using microsurgery. Consequently, patients undergoing DIEP reconstruction have an increased length of hospital stay and increased use of opioid analgesics. According to the Canadian Institute for Health Information, the average hospital cost for a patient undergoing breast reconstruction is $3,715 per day. Reducing postsurgical opioid use and containing healthcare costs is important to the Canadian public and resource-constrained healthcare system.

Enhanced Recovery After Surgery (ERAS) is a multidisciplinary, multimodal, and evidence-based approach to perioperative care that safely reduces hospital length of stay and opioid use following some surgical procedures.16-18 ERAS is the standard of care in colorectal surgery and its advantages are supported by a meta-analysis of 16 randomized controlled trials (RCT). Although ERAS guidelines have been developed for other surgical procedures, the evidence supporting the efficacy of ERAS for non-colorectal surgery is limited. An ERAS guideline for perioperative care of alloplastic and autologous breast reconstruction patients has been established. Main recommendations include minimizing preoperative fasting, postoperative nausea and vomiting prophylaxis, multimodal opioid-sparing analgesia, early feeding and early mobilization. Despite this, the evidence that these recommendations improve care in breast reconstruction is limited. A recent meta-analysis of ERAS in breast reconstruction found that ERAS reduces hospital length of stay by a mean 1.58 days and opioid consumption by 248mg of oral morphine equivalent without an increase in complications. However and to emphasize, none of these studies were RCTs and thus all were subject to the numerous biases associated with observational studies. Currently there is no level-1 evidence to support ERAS in autologous breast reconstruction despite the previously mentioned consensus guideline. A properly designed and executed RCT of ERAS in breast reconstruction would contribute evidence on ERAS in the perioperative care of breast reconstruction patients.

1.3 Objective of the study To conduct a pilot RCT comparing ERAS to conventional perioperative care for patients undergoing autologous DIEP breast reconstruction. As a pilot trial, the primary objective of the study is to assess feasibility outcomes: 1) patient eligibility, 2) recruitment, 3) retention and 4) adherence to the ERAS protocol. The design and conduct of the proposed pilot study will mirror the methodology of the definitive trial including randomization, interventions, and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Women of age 18 years or greater
2. Able to understand and communicate in English
3. Diagnosis of breast cancer or BRCA gene
4. Undergoing (or previously had) unilateral or bilateral mastectomy
5. Undergoing immediate or delayed DIEP breast reconstruction (unilateral or bilateral).

Patients undergoing repeat breast reconstruction (secondary reconstruction) after a previously failed alloplastic or autologous reconstruction will be eligible to participate.

Patients undergoing both DIEP and alloplastic reconstruction (e.g. DIEP reconstruction for one breast, alloplastic reconstruction for the other breast) will also be eligible to participate.

Exclusion Criteria:

1. Non-ambulatory at baseline
2. Pregnant
3. Unable to provide informed consent or unable to complete quality of life questionnaires due to mental capacity, cognitive impairment, or language barrier.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility (pertaining to patient eligibility) | 8-months
  Proportion of screened patients who are eligible for the study
Feasibility (pertaining to patient recruitment) | 8-months
  Proportion of eligible patients who are randomized
Feasibility (pertaining to adherence to follow-up assignment) | 30 days post-surgery
  Proportion of patients with missed assessments and incomplete data variables
Feasibility (pertaining to adherence to ERAS protocol) | Length of inpatient stay (3 to 7+ days)
  Proportion of ERAS interventions followed and achieved

SECONDARY OUTCOMES:
Hospital Length of Stay | 1 week
  Cumulative length of hospital stay post-breast reconstruction.
In-hospital opioid consumption | 1 week
  Cumulative total opioids used during inpatient stay from PACU to discharge converted as oral morphine equivalent. Opioids given during intraoperative phase will not be considered.
BREAST-Q | Preop clinic appointment to 30-days post-surgery
  Reconstruction module of BREAST-Q (patient-reported outcome) obtained at baseline during preoperative clinic visit and 30-days post-surgery.
EQ-5D-5L | Preop clinic appointment to 30-days post-surgery
  General health-related quality of life measure (patient-reported outcome) obtained at baseline during preoperative clinic visit and 30-days post-surgery.
30-days adverse event (composite outcome) | 30-days post-surgery
  Proportion of patients experiencing the following event(s):
  1. Flaps requiring operative salvage or debridement
  2. Hematoma requiring operative drainage/evacuation
  3. Surgical site infection requiring hospital admission and IV antibiotic treatment
  4. DVT
  5. Pulmonary Emboli
  6. Cardiovascular event (myocardial injury, stroke, new atrial fibrillation, congestive heart failure)
30-days additional resource utilization (composite outcome) | 30-days post-surgery
  Proportion of patients requiring:
  1. Visit to ER or Urgent Care
  2. Hospital readmission
  3. Additional surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hyosuk Chin, MD, Principal Investigator — McMaster University; Marko Simunovic, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (2):
- Canada (2):
  - Juravinski Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario